CLINICAL TRIAL: NCT03688256
Title: Obalon Balloon System: Real-World Evidence Commercial Site Registry
Brief Title: Obalon US Commercial Registry
Status: Completed | Type: Observational
Sponsor: Surgical Specialists of Louisiana (Other)
Collaborators: Obalon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 01
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Obalon Balloon System — 6 month Obalon Intragastric Balloons

SUMMARY:
Retrospective study of the data reported in the Obalon US Commercial Registry

DETAILED DESCRIPTION:
Retrospective analyses of the safety and effectiveness data in the Obalon US Commercial Registry reported by participating clinics through August 28, 2018 from patients who started the Obalon therapy from January to December 2017 to represent the first year of commercialization. All patients included in the safety and efficacy analyses must have data through balloon removal and a starting BMI greater than or equal to 25, the definition of overweight and obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Started Obalon Balloon Therapy between Jan.-Dec. 2017
* Weight loss data through balloon removal
* BMI >25kg/m2

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Obalon Commercial Patients
Sampling Method: Non-Probability Sample
Enrollment: 1343 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Primary Safety Outcome - Serious Adverse Events | 6 months
  Percentage of Patients with Serious Adverse Events
Primary Effectiveness Outcome - Weight Loss Metrics | 6 months
  Mean Weight Loss Metrics

IPD SHARING:
Plan to Share IPD: No